CLINICAL TRIAL: NCT05446688
Title: A Phase 2, Multicenter, Non-Randomized, Open-Label, Single-Arm Study to Evaluate the Preliminary Efficacy and Safety of 6MW3211 in Patients With Relapsed or Refractory Lymphoma
Brief Title: A Clinical Study of 6MW3211 Injection in the Treatment of Relapsed/Refractory Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6MW3211-2022-CP201
Record Dates: First submitted 2022-06-27; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6MW3211 (Experimental): 6MW3211 injection, 45mg/kg, Q2W
  Interventions: Drug: 6MW3211

INTERVENTIONS:
Drug: 6MW3211 — 6MW3211 injection, 45mg/kg, Q2W

SUMMARY:
This study is a single arm, non-randomized, open label phase 2 international, multicenter clinical trial to evaluate preliminary efficacy and safety in subjects with relapsed or refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent.
* Age≥18 years.
* Subjects with relapsed or refractory lymphoma.
* Subjects with at least one measurable tumor lesion.
* ECOG 0-2.
* Life expectancy≥3 months.
* Adequate organ functions.

Exclusion Criteria:

* Subjects who had received anticancer therapy or radiotherapy within 21 days or 5 half-lives (whichever is shorter) before enrollment or received adoptive cellular immunotherapy within 12 weeks.
* Subjects who had received allogeneic hematopoietic stem cell transplantation or organ transplantation or received autologous hematopoietic stem cell transplantation within 3 months.
* Subjects with primary or secondary CNS lymphoma.
* History of another malignancy within 3 years before the first dose of investigational drug.
* History of active autoimmune diseases.
* Systemic immunosuppressive therapy within 2 weeks prior to the first dose of investigational drug.
* Subjects who experienced grade 3 or above immune-related adverse events (irAE) .
* Documented history of uncontrolled systemic diseases.
* Subjects who were allergic to any composition of investigational drug.
* Major surgery within 28 days prior to first dose of investigational drug.
* Subjects with active infection.
* Preexisting treatment related toxicity Grade ≥ 2 (except alopecia).
* Subjects with poor treatment compliance.
* Use of any investigational drug or device within 28 days prior to the first dose of investigational drug.
* Live vaccine was administered within 28 days prior to first dose of investigational drug.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 Year
  Defined as the percentage of subjects who experience a best response of either CR or PR

SECONDARY OUTCOMES:
Complete response rate | 1 Year
  Defined as the percentage of subjects who experience a best response of CR
Duration of response | 1 Year
  Time from the date of the first complete response (CR) or partial response (PR) to the earliest date of disease progression or death from any cause
Time to response | 1 Year
  Time from the date of first infusion to the date of confirmed CR or PR
Progression free survival | 1 Year
  Time from the date of first infusion to the earliest date of documented disease progression per radiological evidence or death from any cause
Overall survival | 1 Year
  Time from the date of first infusion until the date of death from any cause
Incidence of adverse events | Up to 28 days post last dose
PK Parameter | 1 Year
  Maximum concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Saijuan Chen, Doctor, Principal Investigator — Ruijin Hospital; Weili Zhao, Doctor, Principal Investigator — Ruijin Hospital